CLINICAL TRIAL: NCT05522478
Title: Effect Of Methylphenidate On Static Balance And Fall Risk In Children With Attention Deficit Hyperactivity Disorder: Cross-Sectional Study
Brief Title: Effect Of Methylphenidate On Balance In Children With Attention Deficit Hyperactivity Disorder
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Gulcan Ozturk
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2022-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; Methylphenidate; Postural Balance
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ADHD group: Children who were diagnosed with ADHD for the first time were classified in the ADHD group (n=33)
  Interventions: Device: Fall risk
- treatment group: children with ADHD who were treated with MPH for a minimum of 3 months were classified in the treatment group (n=32)
  Interventions: Device: Fall risk
- control group: typically developing children were classified in the third-the control group (n=20)
  Interventions: Device: Fall risk

INTERVENTIONS:
Device: Fall risk — Fall risk, static postural balance and sensorimotor integration were assessed using the Biodex Balance System.
  Other Names: static postural balance; sensorimotor integration (m-CTSIB) test

SUMMARY:
Attention Deficit Hyperactivity Disorder is a neurodevelopmental disorder that may have poor motor coordination and balance control. The effect of Methylphenidate treatment on balance and fall risk is still unclear. This study aimed to evaluate the effect of methylphenidate (MPH) treatment on balance, fall risk, and sensorimotor integration in children with Attention Deficit Hyperactivity Disorder (ADHD).

DETAILED DESCRIPTION:
Children who were diagnosed with ADHD for the first time were classified in the ADHD group (n=33), children with ADHD who were treated with MPH for a minimum of 3 months were classified in the treatment group (n=32), and typically developing children were classified in the third-the control group (n=20) in this observational cross-sectional study. Fall risk, static postural balance and sensorimotor integration were assessed using the Biodex Balance System.Postural stability tests, including overall stability index (OSI), anterior-posterior stability index (APSI), and medial-lateral stability index (MLSI), were used to evaluate postural control. The Modified Clinical Test of Sensory Interaction in Balance (m-CTSIB) testing protocol was used to evaluate sensory integration capabilities and balance. Fall risk was evaluated by biodex balance system.

ELIGIBILITY:
Inclusion Criteria:

* Children who were diagnosed with ADHD for the first time according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V, American Psychiatric Association, 2013)

Exclusion Criteria:

* neurological disorders
* psychiatric disorders
* musculoskeletal disorders
* cardiopulmonary diseases
* visual impairments
* developmental coordination disorders that could affect balance

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All children who were diagnosed with ADHD for the first time according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V, American Psychiatric Association, 2013) were classified in the ADHD group (n=33), children with ADHD who were treated with MPH for a minimum of 3 months and were followed-up at our clinic were classified in the treatment group (n=32), and typically developing children were classified in the third-the control group (n=20) in this observational cross-sectional study.
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
postural control | one year
  Postural stability tests, including overall stability index (OSI), anterior-posterior stability index (APSI), and medial-lateral stability index (MLSI)
sensorimotor integration | one year
  The Modified Clinical Test of Sensory Interaction in Balance (m-CTSIB) testing protocol was used to evaluate sensory integration capabilities and balance. Four different conditions were evaluated for the m-CTSIB test protocol: Eyes Open Firm Surface (EOFS), Eyes Closed Firm Surface (ECFS), Eyes Open Soft Surface (EOSS), and Eyes Closed Soft Surface (ECSS)
Fall risk | one year
  Fall risk score was calculated by Biodex balance system

CONTACTS AND LOCATIONS:
Locations (1):
- Gulcan Ozturk, Istanbul, Turkey (Türkiye)